CLINICAL TRIAL: NCT02171364
Title: Clinical Usefulness of Virtual Ablation Guided Catheter Ablation of Atrial Fibrillation: Prospective Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2013-0536
Record Dates: First submitted 2014-06-19; First posted 2014-06-24 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation, Virtual ablation, electrocardiography, electroanatomical mapping data
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- virtual simulation (Experimental): This intervention group is to choose the best effective method operation to patients by simulating 3D atrial computer model which consider patient's heart size and shape.
  Interventions: Procedure: Virtual ablation in based 3D CT of patient who diagnosed AF
- conventional ablation (Active Comparator): The other intervention group is to operate the atrial fibrillation by physician's personal experience, not by virtual simulation.
  Interventions: Procedure: conventional ablation based on physician's personal experience

INTERVENTIONS:
Procedure: Virtual ablation in based 3D CT of patient who diagnosed AF
  Arms: virtual simulation
Procedure: conventional ablation based on physician's personal experience
  Arms: conventional ablation

SUMMARY:
Radiofrequency catheter ablation is highly effective in the treatment of patients with persistent atrial fibrillation. In order to decrease the recurrence rate after catheter ablation, the investigators propose to apply 'virtual' ablation on patient-specific atria by simulating 3D atrial computer model. The investigators will test with five different set of ablation methods and find successful methods for a specific patient. Then, this result will be compared to empirical catheter ablation result by randomly controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AF patients who performed catheter ablation of atrial fibrillation due to uncontrolled pulse rate by anti-arrhythmic drug therapy.

Exclusion Criteria:

* AF patients who have severe heart deformations or blood problems.
* The patients who had been performed catheter ablation of atrial ablation.
* The patients who missed out to recording of 3D CT, echo and electrocardiography.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09-01 (Actual); Study Completion 2015-09-01 (Actual)

PRIMARY OUTCOMES:
change of hospitalization rate | 1, 3, 6, 12, 18 and 24 months after catheter ablation and every 6 months thereafter.

SECONDARY OUTCOMES:
occurence of cardiovascular disease | 6 months
recurrence of AF | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim IS, Lim B, Shim J, Hwang M, Yu HT, Kim TH, Uhm JS, Kim SH, Joung B, On YK, Oh S, Oh YS, Nam GB, Lee MH, Shim EB, Kim YH, Pak HN; CUVIA-AF1 Investigators. Clinical Usefulness of Computational Modeling-Guided Persistent Atrial Fibrillation Ablation: Updated Outcome of Multicenter Randomized Study. Front Physiol. 2019 Dec 17;10:1512. doi: 10.3389/fphys.2019.01512. eCollection 2019. PMID 31920716